CLINICAL TRIAL: NCT01105793
Title: An Open-Label, MultiCenter Evaluation of the Use of Topically Administered FP1198 in Subjects With Pain Associated With Cyclic Mastalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FemmePharma Global Healthcare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP1198-002
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Moderate to Severe Cyclic Mastalgia
Keywords: cyclic mastalgia; cyclic breast pain; fibrocystic breast disease
MeSH Terms: conditions — Fibrocystic Breast Disease | interventions — Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Danazol — High dose FP1198 applied once daily to both breasts for 6 treatment cycles.

SUMMARY:
The purpose of this study is to determine the safety of topical FP1198 for the treatment of moderate to severe cyclic breast pain (cyclic mastalgia) and to examine the clinical activity of FP1198.

ELIGIBILITY:
Inclusion Criteria:

* menstruating females at least 18 years of age
* BMI less than 30
* moderate to severe breast pain associated with the menstrual cycle
* in good general health

Exclusion Criteria:

* pregnant within the last 6 months
* has taken in the last 3 months or currently taking hormonal contraception
* history of malignancy or currently being treated for cancer of the breast or genital organs
* has had breast implants or breast reduction surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Reduction in breast pain | six months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Women's Health Care, San Diego, California
  - Horizons Clinical Research, Denver, Colorado
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Salt Lake Research, Salt Lake City, Utah